CLINICAL TRIAL: NCT00005513
Title: Framingham Nutrition Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5031; R01HL060700 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension

SUMMARY:
To examine hypotheses concerning the relationships between nutrient intake (in particular, specific fatty acids, antioxidant nutrients, and B vitamins), dietary patterns, plasma lipoproteins, and heart disease endpoints in the population-based Framingham Offspring Studies.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Longitudinal analyses were conducted on the associations between diet and cardiovascular and cardiopulmonary disease risk in approximately 3,800 Offspring men and women over eight years of follow-up (from 1984 to present). These analyses considered key nutrients as well as newly defined dietary patterns in Framingham men and women. Cross sectional analyses of diet and plasma lipoprotein relationships in Offspring men and women at two examinations (Exam 3, 1984-88; and Exam 5, 1991-94) were also conducted. All analyses evaluated the total (direct and indirect) and joint effects of dietary nutrients. Where appropriate, analyses controlled for plasma nutrient levels (folacin, vitamins B6 and B12 and homocysteine). The influence of potential confounding variables, effect modifiers, and intervening variables that lie in the causal pathway were examined, as appropriate to the statistical model, including traditional cardiovascular disease risk factors and apoE isoform status.

Several existing Framingham data sets were utilized, including comprehensive data sets on nutrient intake, cardiovascular disease risk factors, clinically verified cardiovascular and cardiopulmonary endpoints and other covariates. The Offspring Exam 3 and 5 nutrition data sets included multiple day assessments of dietary intake which improved the ability to detect relationships of interest. The investigators completed the Framingham Food Habit Questionnaire data set for Exam 5; this instrument included important covariates for the analyses (including vitamin supplement use).

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Millen — Boston University

REFERENCES:
- [Background] Millen BE, Quatromoni PA, Copenhafer DL, Demissie S, O'Horo CE, D'Agostino RB. Validation of a dietary pattern approach for evaluating nutritional risk: the Framingham Nutrition Studies. J Am Diet Assoc. 2001 Feb;101(2):187-94. doi: 10.1016/s0002-8223(01)00051-7. PMID 11271691
- [Background] Millen BE, Quatromoni PA. Nutritional research within the Framingham Heart Study. J Nutr Health Aging. 2001;5(3):139-43. PMID 11458282
- [Background] Quatromoni PA, Copenhafer DL, Demissie S, D'Agostino RB, O'Horo CE, Nam BH, Millen BE. The internal validity of a dietary pattern analysis. The Framingham Nutrition Studies. J Epidemiol Community Health. 2002 May;56(5):381-8. doi: 10.1136/jech.56.5.381. PMID 11964437
- [Background] Millen BE, Quatromoni PA, Nam BH, O'Horo CE, Polak JF, D'Agostino RB. Dietary patterns and the odds of carotid atherosclerosis in women: the Framingham Nutrition Studies. Prev Med. 2002 Dec;35(6):540-7. doi: 10.1006/pmed.2002.1116. PMID 12460521